CLINICAL TRIAL: NCT03447314
Title: A Phase I, Open-Label Study of GSK1795091 Administered in Combination With Immunotherapies in Participants With Advanced Solid Tumors
Brief Title: Study of a Combination of GSK1795091 and Immunotherapies in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 204686; 2017-003545-23 (EudraCT Number)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Neoplasms
Keywords: pembrolizumab; GSK1795091; Dose-escalation; 204686; Immunotherapies; GSK3359609; Phase I; anticancer agent; OX40; 201212; 204691; ICOS; TLR4; GSK3174998; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — TLR4 agonist GSK1795091; pembrolizumab

STUDY DESIGN:
Intervention Model Description: In Part 1, one dose level of GSK3174998, GSK3359609, or pembrolizumab with up to 5 dose levels of GSK1795091 are planned for evaluation. Sequential cohorts will be enrolled and dose escalation (or de-escalation) will proceed according to Neuenschwander-Continual Reassessment Method (N-CRM design). In Part 2, subjects will be administered GSK1795091 in combination with either 24 mg GSK3174998, 80 mg GSK3359609, or 200 mg pembrolizumab at a dose identified in Part 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Part 1a: 50ng GSK1795091 + 24mg GSK3174998 (Experimental): Participants will be administered GSK1795091 50 nanogram (ng) intravenously (IV) on Days 1 and 8 followed by once weekly administration of GSK1795091 50 ng IV in combination with GSK3174998 24 milligram (mg) administered at 3-week intervals (Q3W) via the IV route until Week 12. From Week 12 onwards, GSK1795091 50 ng IV will be administered in combination with GSK3174998 24 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3174998
- Part 1a: 100ng GSK1795091 + 24mg GSK3174998 (Experimental): Participants will be administered GSK1795091 100 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 100 ng IV in combination with GSK3174998 24 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 100 ng IV will be administered in combination with GSK3174998 24 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3174998
- Part 1a: 150ng GSK1795091 + 24mg GSK3174998 (Experimental): Participants will be administered GSK1795091 150 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 150 ng IV in combination with GSK3174998 24 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 150 ng IV will be administered in combination with GSK3174998 24 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3174998
- Part 1a: 200ng GSK1795091 + 24mg GSK3174998 (Experimental): Participants will be administered GSK1795091 200 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 200 ng IV in combination with GSK3174998 24 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 200 ng IV will be administered in combination with GSK3174998 24 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3174998
- Part 1a: 250ng GSK1795091 + 24mg GSK3174998 (Experimental): Participants will be administered GSK1795091 250 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 250 ng IV in combination with GSK3174998 24 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 250 ng IV will be administered in combination with GSK3174998 24 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3174998
- Part 1b: 50ng GSK1795091 + 80mg GSK3359609 (Experimental): Participants will be administered GSK1795091 50 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 50 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 50 ng IV will be administered in combination with GSK3359609 80 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3359609
- Part 1b: 100ng GSK1795091 + 80mg GSK3359609 (Experimental): Participants will be administered GSK1795091 100 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 100 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 100 ng IV will be administered in combination with GSK3359609 80 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3359609; Drug: Pembrolizumab
- Part 1b: 150ng GSK1795091 + 80mg GSK3359609 (Experimental): Participants will be administered GSK1795091 150 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 150 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 150 ng IV will be administered in combination with GSK3359609 80 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3359609
- Part 1b: 200ng GSK1795091 + 80mg GSK3359609 (Experimental): Participants will be administered GSK1795091 200 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 200 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 200 ng IV will be administered in combination with GSK3359609 80 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3359609
- Part 1b: 250ng GSK1795091 + 80mg GSK3359609 (Experimental): Participants will be administered GSK1795091 250 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 250 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 250 ng IV will be administered in combination with GSK3359609 80 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: GSK3359609
- Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab (Experimental): Participants will be administered GSK1795091 50 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 50 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 50 ng IV will be administered in combination with pembrolizumab 200 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: Pembrolizumab
- Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab (Experimental): Participants will be administered GSK1795091 100 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 100 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 100 ng IV will be administered in combination with pembrolizumab 200 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: Pembrolizumab
- Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab (Experimental): Participants will be administered GSK1795091 150 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 150 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 150 ng IV will be administered in combination with pembrolizumab 200 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: Pembrolizumab
- Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab (Experimental): Participants will be administered GSK1795091 200 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 200 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 200 ng IV will be administered in combination with pembrolizumab 200 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: Pembrolizumab
- Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab (Experimental): Participants will be administered GSK1795091 250 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 250 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 250 ng IV will be administered in combination with pembrolizumab 200 mg at Q3W interval.
  Interventions: Drug: GSK1795091; Drug: Pembrolizumab
- Part 2a: GSK1795091 + 24 mg GSK3174998 (Experimental): Participants will be administered GSK1795091 at a dose identified in Part 1 along with GSK3174998 24 mg.
  Interventions: Drug: GSK1795091; Drug: GSK3174998
- Part 2b: GSK1795091 + 80 mg GSK3359609 (Experimental): Participants will be administered GSK1795091 at a dose identified in Part 1 along with GSK3359609 80 mg.
  Interventions: Drug: GSK1795091; Drug: GSK3359609
- Part 2c: GSK1795091 + 200 mg Pembrolizumab (Experimental): Participants will be administered GSK1795091 at a dose identified in Part 1 along with pembrolizumab 200 mg.
  Interventions: Drug: GSK1795091; Drug: Pembrolizumab

INTERVENTIONS:
Drug: GSK1795091 — GSK1795091 will be available as solution for injection
Drug: GSK3174998 — GSK3174998 will be available as lyophilized powder to be reconstituted for infusion.
  Arms: Part 1a: 100ng GSK1795091 + 24mg GSK3174998; Part 1a: 150ng GSK1795091 + 24mg GSK3174998; Part 1a: 200ng GSK1795091 + 24mg GSK3174998; Part 1a: 250ng GSK1795091 + 24mg GSK3174998; Part 1a: 50ng GSK1795091 + 24mg GSK3174998; Part 2a: GSK1795091 + 24 mg GSK3174998
Drug: GSK3359609 — GSK3359609 will be available as solution for infusion.
  Arms: Part 1b: 100ng GSK1795091 + 80mg GSK3359609; Part 1b: 150ng GSK1795091 + 80mg GSK3359609; Part 1b: 200ng GSK1795091 + 80mg GSK3359609; Part 1b: 250ng GSK1795091 + 80mg GSK3359609; Part 1b: 50ng GSK1795091 + 80mg GSK3359609; Part 2b: GSK1795091 + 80 mg GSK3359609
Drug: Pembrolizumab — Pembrolizumab will be available as solution for infusion or lyophilized powder for reconstitution.
  Arms: Part 1b: 100ng GSK1795091 + 80mg GSK3359609; Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab; Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab; Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab; Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab; Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab; Part 2c: GSK1795091 + 200 mg Pembrolizumab

SUMMARY:
GSK1795091 is being developed for administration in combination with other immune system modulators for the treatment of cancers. The study will be conducted in two parts. In Part 1, dose escalation will be performed to identify combination dose levels comprising GSK1795091 with either 24 milligrams (mg) GSK3174998 (Part 1a), 80 mg GSK3359609 (Part 1b), or 200 mg pembrolizumab (Part 1c). One dose level of GSK3174998, GSK3359609, or pembrolizumab with up to 5 dose levels of GSK1795091 are planned for evaluation. In Part 2 (dose-expansion), subjects will receive a single dose level of GSK1795091 as identified based on data from Part 1, in combination with either GSK3174998, GSK3359609, or pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be >=18 years of at the time of signing the informed consent.
* Histological documentation of advanced solid tumor.
* Archival tumor tissue obtained at any time from the initial diagnosis to study entry. Although a fresh biopsy obtained during screening is preferred, archival tumor specimen is acceptable if it is not feasible to obtain a fresh biopsy. Subjects enrolled in a PK/Pharmacodynamic Cohort must provide a fresh biopsy of a tumor lesion not previously irradiated during the screening period and must agree to provide at least one additional on-treatment biopsy.
* Disease that has progressed after standard therapies or for which standard therapy is otherwise unsuitable (example, intolerance).
* Measurable disease, that is, presenting with at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Life expectancy of at least 12 weeks.
* Adequate organ function.
* In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.
* Male or female subjects will be included. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: a) Not a woman of childbearing potential (WOCBP) OR b). A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions specified.

Additional Inclusion criteria for Subjects in Part 2a (GSK3174998 expansion) and Part 2b (GSK3359609 expansion):

* Histological or cytological documentation of squamous cell carcinoma of the head and neck (SCCHN) (oral cavity, oropharynx, hypopharynx, or larynx) that is recurrent, locally advanced, or metastatic and is not amenable to curative treatment options, surgery or definitive chemoradiation therapy.
* Received, ineligible for, or otherwise unsuitable for platinum-based therapy and anti-Programmed death receptor-1 (PD-1)/programmed death-ligand 1 (PD-L1) therapy
* Received no more than 3 prior lines of systemic therapy for metastatic disease.

Additional Inclusion Criteria for Subjects in Part 2c (pembrolizumab expansion):

* Histological or cytological documentation of SCCHN (oral cavity, oropharynx, hypopharynx, or larynx) that is recurrent, locally advanced, or metastatic and is not amenable to curative treatment options, surgery or definitive chemoradiation therapy.
* Received no more than 2 prior lines of systemic therapy for metastatic disease.

Exclusion Criteria:

* Malignancy other than disease under study with the exception of those from which the subject has been disease-free for more than 2 years and not expected to affect the safety of the subject or the endpoints of the trial.
* Symptomatic central nervous system (CNS) metastases or asymptomatic CNS metastases that have required steroids within 2 weeks prior to first dose of study treatment.
* Active autoimmune disease that has required systemic disease modifying or immunosuppressive treatment within the last 2 years. Replacement therapy (example, thyroxine or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted.
* Concurrent medical condition requiring the use of systemic immunosuppressive treatment within 28 days before the first dose of study treatment.
* Known human immunodeficiency virus infection.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study treatment.
* Positive Hepatitis C test result at screening or within 3 months prior to first dose of study treatment.
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 milliseconds (msec) or QTcF >480 msec for subjects with bundle branch block
* Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction.
* Recent history of allergen desensitization therapy within 4 weeks of starting study treatment.
* History of severe hypersensitivity to monoclonal antibodies (mAbs).
* History or evidence of cardiovascular (CV) risk including any of the following: a) Recent (within the past 6 months) history of serious uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities including second degree (Type II) or third degree atrioventricular block. b) Cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting within the past 6 months before enrollment. c) Congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association (NYHA) functional classification system. d) Recent (within the past 6 months) history of symptomatic pericarditis.
* History of idiopathic pulmonary fibrosis, pneumonitis, interstitial lung disease, or organizing pneumonia, or evidence of active, non-infectious pneumonitis.
* Recent history (within 6 months) of uncontrolled symptomatic ascites or pleural effusions.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other condition that could interfere with the subject's safety, obtaining informed consent, or compliance to the study procedures.
* Is or has an immediate family member (example, spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective Institutional Review Board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
* Prior treatment with the following agents: a) OX40, inducible T-cell co-stimulator (ICOS) agonist at any time. b) Prior systemic or intratumoral therapy with TLR agonist. c) Anticancer therapy or investigational therapy within 30 days or 5 half-lives of the drug, whichever is shorter. d) Prior radiation therapy: permissible if at least 1 non-irradiated measurable lesion is available for assessment according to RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. A wash out of at least 14 days before start of study treatment for radiation of any intended use to the extremities for bone metastases and 28 days for radiation to the chest, brain, or visceral organs is required.
* Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.
* Toxicity from previous treatment including: a) Toxicity Grade >=3 related to prior immunotherapy and that lead to study treatment discontinuation. b) Toxicity related to prior treatment has not resolved to Grade <=1 (except alopecia, or endocrinopathy managed with replacement therapy).
* Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor, and recombinant erythropoietin) within 2 weeks before the first dose of study treatment.
* Major surgery <=4 weeks before the first dose of study treatment. Subjects must have also fully recovered from any surgery (major or minor) and/or its complications before initiating study treatment.
* Known drug or alcohol abuse.
* Receipt of any live vaccine within 4 weeks.

Additional Exclusion Criteria for Subjects in Part 2c

* Received prior anti-PD-1/PD-L1 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (5):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Tacoma, Washington
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Amsterdam, Netherlands
- GSK Investigational Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Derived] Steeghs N, Hansen AR, Hanna GJ, Garralda E, Park H, Strauss J, Adam M, Campbell G, Carver J, Easton R, Mays K, Skrdla P, Struemper H, Washburn ML, Matheny C, Piha-Paul SA. Manufacturing-dependent change in biological activity of the TLR4 agonist GSK1795091 and implications for lipid A analog development. Clin Transl Sci. 2022 Nov;15(11):2625-2639. doi: 10.1111/cts.13387. Epub 2022 Sep 12. PMID 36097345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomized, open-label study of GSK1795091 administered in combination with immunotherapies in participants with advanced solid tumors.
Pre-assignment Details: Total 54 participants were enrolled in the study. GSK1795091 150 nanograms (ng), 200 and 250 ng arms of Parts 1b and 1c were not initiated as GSK1795091 was no longer supplied due to manufacturing issue. Part 2 was not initiated.
Groups:
- Part 1a: 50ng GSK1795091 + 24mg GSK3174998: Participants were administered GSK1795091 50 ng intravenously (IV) on Days 1 and 8 followed by once weekly administration of GSK1795091 50 ng IV in combination with GSK3174998 24 milligram (mg) administered at 3-week intervals (Q3W) via the IV route until Week 12. From Week 12 onwards, GSK1795091 50 ng IV was administered in combination with GSK3174998 24 mg at Q3W interval.
- Part 1a: 100ng GSK1795091 + 24mg GSK3174998: Participants were administered GSK1795091 100 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 100 ng IV in combination with GSK3174998 24 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 100 ng IV was administered in combination with GSK3174998 24 mg at Q3W interval.
- Part 1a: 150ng GSK1795091 + 24mg GSK3174998: Participants were administered GSK1795091 150 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 150 ng IV in combination with GSK3174998 24 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 150 ng IV was administered in combination with GSK3174998 24 mg at Q3W interval.
- Part 1a: 200ng GSK1795091 + 24mg GSK3174998: Participants were administered GSK1795091 200 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 200 ng IV in combination with GSK3174998 24 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 200 ng IV was administered in combination with GSK3174998 24 mg at Q3W interval.
- Part 1a: 250ng GSK1795091 + 24mg GSK3174998: Participants were administered GSK1795091 250 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 250 ng IV in combination with GSK3174998 24 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 250 ng IV was administered in combination with GSK3174998 24 mg at Q3W interval.
- Part 1b: 50ng GSK1795091 + 80mg GSK3359609: Participants were administered GSK1795091 50 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 50 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 50 ng IV was administered in combination with GSK3359609 80 mg at Q3W interval.
- Part 1b: 100ng GSK1795091 + 80mg GSK3359609: Participants were administered GSK1795091 100 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 100 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 100 ng IV was administered in combination with GSK3359609 80 mg at Q3W interval.
- Part 1b: 150ng GSK1795091 + 80mg GSK3359609: Participants were planned to administer GSK1795091 150 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 150 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 150 ng IV was planned to administer in combination with GSK3359609 80 mg at Q3W interval.
- Part 1b: 200ng GSK1795091 + 80mg GSK3359609: Participants were planned to administer GSK1795091 200 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 200 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 200 ng IV was planned to administer in combination with GSK3359609 80 mg at Q3W interval.
- Part 1b: 250ng GSK1795091 + 80mg GSK3359609: Participants were planned to administer GSK1795091 250 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 250 ng IV in combination with GSK3359609 80 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 250 ng IV was planned to administer in combination with GSK3359609 80 mg at Q3W interval.
- Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab: Participants were administered GSK1795091 50 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 50 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 50 ng IV was administered in combination with pembrolizumab 200 mg at Q3W interval.
- Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab: Participants were administered GSK1795091 100 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 100 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 100 ng IV was administered in combination with pembrolizumab 200 mg at Q3W interval.
- Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab: Participants were planned to administer GSK1795091 150 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 150 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 150 ng IV was planned to administer in combination with pembrolizumab 200 mg at Q3W interval.
- Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab: Participants were planned to administer GSK1795091 200 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 200 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 200 ng IV was planned to administer in combination with pembrolizumab 200 mg at Q3W interval.
- Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab: Participants were planned to administer GSK1795091 250 ng IV on Days 1 and 8 followed by once weekly administration of GSK1795091 250 ng IV in combination with pembrolizumab 200 mg administered at Q3W via the IV route until Week 12. From Week 12 onwards, GSK1795091 250 ng IV was planned to administer in combination with pembrolizumab 200 mg at Q3W interval.
- Part 2a: GSK1795091 + 24 mg GSK3174998: Participants were planned to receive GSK1795091 at a dose identified in Part 1 along with GSK3174998 24 mg.
- Part 2b: GSK1795091 + 80 mg GSK3359609: Participants were planned to receive GSK1795091 at a dose identified in Part 1 along with GSK3359609 80 mg.
- Part 2c: GSK1795091 + 200 mg Pembrolizumab: Participants were planned to receive GSK1795091 at a dose identified in Part 1 along with pembrolizumab 200 mg.
Period: Part 1 (Up to 47 Months and 13 Days)
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Started | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 5 | 7 | 4 | 1 | 6 | 3 | 0 | 0 | 0 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 6 | 5 | 4 | 3 | 1 | 4 | 2 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason for discontinuation was not recorded in the case report form | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator discretion | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Up to 47 Months and 13 Days)
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 1b and Part 1c (GSK1795091 150ng, 200ng, 250ng arms) were not initiated as GSK1795091 was no longer supplied due to a manufacturing issue. Hence, no participants were enrolled in Part 1b and Part 1c (GSK1795091 150ng, 200ng, 250ng arms); Part 2 was not initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab | Total
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 54
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  19 - 64 years | 8 | 3 | 7 | 3 | 0 | 5 | 4 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 37
  >=65 years | 1 | 3 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 2 | 0 | 4 | 3 | 0 | 0 | 0 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 28
  Male | 5 | 3 | 6 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian - Central/South Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White - Arabic/North African Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White - White/Caucasian/European Heritage | 6 | 6 | 7 | 4 | 2 | 5 | 5 | 0 | 0 | 0 | 6 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 46
  Unknown | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs (STEAEs)
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A serious adverse event is defined as any untoward medical occurrence that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement or associated with liver injury and impaired liver function. TEAEs are defined as adverse events that started or worsened in severity on or after the first dose of study medication. All Treated Population consisted of all participants who received at least 1 dose of GSK1795091, GSK3174998, GSK3359609, or pembrolizumab.
Time Frame: Up to 27 months
Population: All Treated Population. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Parts 1b and 1c as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  TEAEs | 9 | 6 | 9 | 4 | 1 | 6 | 5 |  |  |  | 5 | 6 |  |  |
  STEAEs | 1 | 2 | 5 | 1 | 0 | 2 | 2 |  |  |  | 3 | 2 |  |  |

2. Primary Outcome: Part 2: Number of Participants With TEAEs and STEAEs
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A serious adverse event is defined as any untoward medical occurrence that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement or associated with liver injury and impaired liver function. TEAEs are defined as adverse events that started or worsened in severity on or after the first dose of study medication.
Time Frame: Up to 27 months
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Dose-limiting Toxicity (DLT)
Description: An adverse event was considered to be a DLT if it was considered by investigator to be clinically relevant and attributed (definitely, probably or possibly) to study treatment and met one of the criteria: hematologic toxicity-Grade4 neutropenia of >7 days duration or febrile neutropenia, Grade 4 anemia, Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding as described in Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, non-hematologic toxicity-Grade 4 toxicity, Grade 3 toxicity that does not resolve to <=Grade 1 or Baseline within 14 days despite optimal supportive care, alanine aminotransferase (ALT) >=5 times upper limit of normal (ULN), ALT >=3 times ULN persists for >=4 weeks, ALT >=3 times ULN and bilirubin >=2 times ULN (>35 percent [%] direct bilirubin), ALT >=3 times ULN and international normalized ratio (INR) >1.5, ALT >=3 times ULN associated with symptoms (new or worsening) believed to be related to liver injury or hypersensitivity.
Time Frame: 42 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 |  |  |  | 0 | 1 |  |  |

4. Primary Outcome: Part 1: Number of Participants With TEAEs Leading to Discontinuation
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. TEAEs are defined as adverse events that started or worsened in severity on or after the first dose of study medication.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 1 |  |  |  | 0 | 1 |  |  |

5. Primary Outcome: Part 2: Number of Participants With TEAEs Leading to Discontinuation
Description: as for outcome 4
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: Part 1: Number of Participants With TEAEs Leading to Dose Reductions or Dose Delays
Description: as for outcome 4
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants | 4 | 2 | 1 | 1 | 0 | 2 | 2 |  |  |  | 4 | 2 |  |  |

7. Primary Outcome: Part 2: Number of Participants With TEAEs Leading to Dose Reductions or Dose Delays
Description: as for outcome 4
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: Part 1: Number of Participants With Change From Baseline in Hematology Parameters With Respect to the Normal Range
Description: Blood samples were collected for the analysis of following hematology parameters: neutrophils (Neutro), lymphocytes (lympho), monocytes (Mono), eosinophils (Eosino), basophils (Baso), hemoglobin (Hb), hematocrit (Hct), erythrocytes (Erythro), erythrocyte mean corpuscular volume (EMCV), erythrocyte mean corpuscular hemoglobin (EMCH) and platelet count (PC). Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Data was categorized as decrease to low (D to L) (value below lower limit of normal range [LNR]) and increase to high (I to H) (value above upper LNR). Participants were counted twice if participant had both decreased to low and increased to high within an assessment. Data for worst-case on therapy for categories decrease to low and increase to high is presented.
Time Frame: Baseline (Day 1: Pre-dose) and up to 2 years
Population: All Treated Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles). Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Parts 1b and 1c as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  Neutro, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Neutro, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 1 |  |  |
  Neutro, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Neutro, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 0 | 1 | 1 | 0 | 1 | 1 |  |  |  | 3 | 2 |  |  |
  Lympho, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Lympho, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 4 | 1 | 3 | 0 | 0 | 4 | 0 |  |  |  | 1 | 1 |  |  |
  Lympho, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Lympho, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 1 |  |  |
  Mono, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Mono, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  Mono, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Mono, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 |  |  |  | 0 | 3 |  |  |
  Eosino, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Eosino, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 |  |  |  | 0 | 1 |  |  |
  Eosino, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Eosino, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 |  |  |  | 0 | 2 |  |  |
  Baso, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Baso, D to L, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  Baso, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Baso, I to H, n=8,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  Hb, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 |  |  |  | 2 | 0 |  |  |
  Hb, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  Hct, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 0 | 3 | 1 | 0 | 3 | 1 |  |  |  | 4 | 2 |  |  |
  Hct, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  Erythro, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 2 | 2 | 1 | 0 | 1 | 2 |  |  |  | 2 | 2 |  |  |
  Erythro, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  EMCV, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 2 | 3 | 0 | 0 | 1 | 1 |  |  |  | 2 | 0 |  |  |
  EMCV, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 |  |  |  | 0 | 0 |  |  |
  EMCH, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 1 | 4 | 1 | 0 | 2 | 2 |  |  |  | 2 | 2 |  |  |
  EMCH, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 |  |  |  | 0 | 0 |  |  |
  PC, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  PC, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 |  |  |  | 1 | 3 |  |  |

9. Primary Outcome: Part 2: Number of Participants With Change From Baseline in Hematology Parameters With Respect to the Normal Range
Description: Blood samples were planned to be collected for the analysis of following hematology parameters: neutrophils, lymphocytes, monocytes, eosinophils, basophils, hemoglobin, hematocrit, erythrocytes, erythrocyte mean corpuscular volume, erythrocyte mean corpuscular hemoglobin and platelet count.
Time Frame: Baseline (Day 1: Pre-dose) and up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Part 1: Number of Participants With Change From Baseline in Chemistry Parameters With Respect to the Normal Range
Description: Blood samples were collected for the analysis of following chemistry parameters: urea, creatinine (Cr), glucose (Glu), potassium (Pot), sodium (Sod), calcium (Cal), aspartate aminotransferase (AST), ALT, alkaline phosphatase (ALP), bilirubin (Bil), direct bilirubin (D.Bil), protein, albumin (Alb), C-reactive protein (CRP) and Creatinine Clearance (CrCl). Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Data was categorized as decrease to low (value below the lower LNR), and increase to high (value above the upper LNR). Participants were counted twice if the participant had both decreased to low and increased to high within an assessment. Data for worst case on therapy for categories decrease to low and increase to high is presented.
Time Frame: Baseline (Day 1: Pre-dose) and up to 2 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  Urea, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 |  |  |  | 1 | 1 |  |  |
  Urea, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 1 | 1 | 1 | 0 | 2 | 0 |  |  |  | 0 | 2 |  |  |
  Cr, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 |  |  |  | 4 | 1 |  |  |
  Cr, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 4 | 2 | 0 | 1 | 0 | 1 | 1 |  |  |  | 0 | 0 |  |  |
  Glu, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |  |  |  | 0 | 1 |  |  |
  Glu, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 0 | 1 | 2 | 1 | 2 | 1 |  |  |  | 1 | 2 |  |  |
  Pot, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1 | 2 |  |  |
  Pot, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 |  |  |  | 0 | 1 |  |  |
  Sod, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 1 | 2 | 1 | 0 | 2 | 1 |  |  |  | 3 | 2 |  |  |
  Sod, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  Cal, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 |  |  |  | 2 | 0 |  |  |
  Cal, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 |  |  |  | 1 | 1 |  |  |
  AST, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  AST, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 2 | 2 | 2 | 0 | 2 | 0 |  |  |  | 2 | 1 |  |  |
  ALT, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  ALT, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 1 | 3 | 2 | 0 | 3 | 1 |  |  |  | 0 | 1 |  |  |
  ALP, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  ALP, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 1 | 2 | 1 | 0 | 0 | 1 |  |  |  | 2 | 0 |  |  |
  Bil, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  | 0 | 1 |  |  |
  Bil, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 |  |  |  | 2 | 0 |  |  |
  D.Bil, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  D.Bil, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 |  |  |  | 1 | 0 |  |  |
  Protein, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 0 | 1 | 2 | 0 | 2 | 0 |  |  |  | 3 | 1 |  |  |
  Protein, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  | 0 | 1 |  |  |
  Alb, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 2 | 2 | 2 | 0 | 1 | 0 |  |  |  | 1 | 2 |  |  |
  Alb, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  CRP, D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  CRP, I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 1 | 2 | 0 | 1 | 1 | 0 |  |  |  | 1 | 1 |  |  |
  CrCl, D to L, n=1,2,3,1,1,4,0,0,0,0,1,2,0,0,0: number analyzed (Participants) | 1 | 2 | 3 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  CrCl, D to L, n=1,2,3,1,1,4,0,0,0,0,1,2,0,0,0 | 0 | 0 | 2 | 0 | 0 | 0 |  |  |  |  | 0 | 0 |  |  |
  CrCl, I to H, n=1,2,3,1,1,4,0,0,0,0,1,2,0,0,0: number analyzed (Participants) | 1 | 2 | 3 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  CrCl, I to H, n=1,2,3,1,1,4,0,0,0,0,1,2,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0 | 0 |  |  |

11. Primary Outcome: Part 2: Number of Participants With Change From Baseline in Chemistry Parameters With Respect to the Normal Range
Description: Blood samples were planned to be collected for the analysis of following chemistry parameters: urea, creatinine, glucose, potassium, sodium, calcium, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, bilirubin, direct bilirubin, protein, albumin, C-reactive protein and Creatinine Clearance.
Time Frame: Baseline (Day 1: Pre-dose) and up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

12. Primary Outcome: Part 1: Number of Participants With Worst Case Urinalysis Results Relative to Normal Range Criteria
Description: Urine samples were collected for the analysis of following urinalysis parameters: glucose (Glu), protein (Pro), occult blood (OB), ketones, potential of hydrogen (pH) and specific gravity (SpGr) by dipstick method. The dipstick test gives results in a semi-quantitative manner. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The reference range is 1.002-1.030. Urine pH is an acid-base measurement. Normal urine has a slightly acid pH (5.0 - 6.0). Data was categorized as decrease to low (value below the lower LNR) and increase to high (value above the upper LNR). Participants were counted twice if the participant had both decreased to low and increased to high within an assessment. Data for worst-case on therapy for categories decrease to low and increase to high is presented.
Time Frame: Up to 2 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  Glu: D to L, n=9,5,8,1,2,4,2,0,0,0,0,5,0,0,0: number analyzed (Participants) | 9 | 5 | 8 | 1 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  Glu: D to L, n=9,5,8,1,2,4,2,0,0,0,0,5,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0 |  |  |
  Glu: I to H, n=9,5,8,1,2,4,2,0,0,0,0,5,0,0,0: number analyzed (Participants) | 9 | 5 | 8 | 1 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  Glu: I to H, n=9,5,8,1,2,4,2,0,0,0,0,5,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0 |  |  |
  Pro: D to L, n=9,2,7,1,2,4,0,0,0,0,4,0,0,0,0: number analyzed (Participants) | 9 | 2 | 7 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
  Pro: D to L, n=9,2,7,1,2,4,0,0,0,0,4,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0 |  |  |  |
  Pro: I to H, n=9,2,7,1,2,4,0,0,0,0,4,0,0,0,0: number analyzed (Participants) | 9 | 2 | 7 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
  Pro: I to H, n=9,2,7,1,2,4,0,0,0,0,4,0,0,0,0 | 3 | 0 | 2 | 0 | 0 | 0 |  |  |  |  | 0 |  |  |  |
  OB: D to L, n=4,5,8,1,1,4,2,0,0,0,1,4,0,0,0: number analyzed (Participants) | 4 | 5 | 8 | 1 | 1 | 4 | 2 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0
  OB: D to L, n=4,5,8,1,1,4,2,0,0,0,1,4,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  OB: I to H, n=4,5,8,1,1,4,2,0,0,0,1,4,0,0,0: number analyzed (Participants) | 4 | 5 | 8 | 1 | 1 | 4 | 2 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0
  OB: I to H, n=4,5,8,1,1,4,2,0,0,0,1,4,0,0,0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  Ketones: D to L, n=9,5,8,1,2,4,2,0,0,0,0,5,0,0,0: number analyzed (Participants) | 9 | 5 | 8 | 1 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  Ketones: D to L, n=9,5,8,1,2,4,2,0,0,0,0,5,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  | 0 |  |  |
  Ketones: I to H, n=9,5,8,1,2,4,2,0,0,0,0,5,0,0,0: number analyzed (Participants) | 9 | 5 | 8 | 1 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  Ketones: I to H, n=9,5,8,1,2,4,2,0,0,0,0,5,0,0,0 | 3 | 0 | 3 | 1 | 0 | 1 | 1 |  |  |  |  | 0 |  |  |
  pH: D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  pH: I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 |  |  |  | 1 | 1 |  |  |
  SpGr: D to L, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  SpGr: I to H, n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 |  |  |  | 1 | 0 |  |  |

13. Primary Outcome: Part 2: Number of Participants With Worst Case Urinalysis Results Relative to Normal Range Criteria
Description: Urine samples were planned to be collected for the analysis of following urine parameters: glucose, protein, occult blood, ketones, potential of hydrogen and specific gravity by dipstick method.
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

14. Primary Outcome: Part 1: Number of Participants With Increase From Baseline in Vital Signs According to Markedly Abnormal Criteria
Description: Vital signs including systolic blood pressure (SBP), diastolic BP (DBP), pulse rate (PR) and body temperature (BT) were measured in a semi-supine position after 5 minutes rest for the participants. SBP: Category1 (>140 and <161 millimeter of mercury[mmHg]), Category 2 (>=161 and <181 mmHg), Category3 (>=181 mmHg); DBP: Category1 (>90 and <101 mmHg), Category 2 (>=101 and <111 mmHg), Category 3 (>=111 mmHg); PR: Category 1 (>101 and <116 beats per minutes[bpm]), Category 2 (>=116 and <131 bpm), Category 3 (>=131 bpm); BT: Category 1 (>38.0 and <38.6 degrees Celsius), Category 2 (>=38.6 and <39.1 degrees Celsius), Category 3 (>=39.1 degrees Celsius). Data for any increase in category at worst case on therapy is presented.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  Any increase, SBP | 7 | 3 | 6 | 3 | 1 | 1 | 2 |  |  |  | 2 | 3 |  |  |
  Any increase, DBP | 1 | 1 | 3 | 1 | 1 | 1 | 0 |  |  |  | 0 | 3 |  |  |
  Any increase, Pulse rate | 2 | 1 | 4 | 1 | 0 | 1 | 2 |  |  |  | 1 | 2 |  |  |
  Any increase, Body temperature | 1 | 1 | 2 | 1 | 0 | 0 | 0 |  |  |  | 1 | 0 |  |  |

15. Primary Outcome: Part 2: Number of Participants With Vital Signs Any Increases From Baseline According to Markedly Abnormal Criteria
Description: Vital signs including SBP, DBP, pulse rate and body temperature were planned to be measured in a semi-supine position after 5 minutes rest for the participants.
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

16. Primary Outcome: Part 1: Number of Participants With Any Decrease From Baseline in Vital Sign According to Markedly Abnormal Criteria
Description: Vital signs including SBP, DBP and pulse rate were measured in a semi-supine position after 5 minutes rest for the participants. For SBP: a decrease in Category was defined as <80 mmHg decrease from Baseline; DBP: decrease defined as Category (<50 mmHg decrease from Baseline); pulse rate: decrease defined as Category (<45 bpm decrease from Baseline). Data for decrease in category at worst case on therapy is presented.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  Any decrease, SBP | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 0 |  |  |
  Any decrease, DBP | 2 | 1 | 1 | 0 | 0 | 1 | 0 |  |  |  | 0 | 0 |  |  |
  Any decrease, Pulse rate | 0 | 0 | 0 | 1 | 0 | 1 | 0 |  |  |  | 0 | 0 |  |  |

17. Primary Outcome: Part 2: Number of Participants With Vital Signs Any Decreases From Baseline According to Markedly Abnormal Criteria
Description: Vital signs including SBP, DBP and pulse rate were planned to be measured in a semi-supine position after 5 minutes rest for the participants.
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

18. Primary Outcome: Part 1: Number of Participants With Any Increase From Baseline in Corrected QT Interval Using Fredericia's Formula (QTcF) According to Markedly Abnormal Criteria
Description: 12-lead electrocardiogram (ECG) was obtained at indicated time point using an automated ECG machine that measured QTcF interval. QTc parameters were graded according to National Cancer Institute - CTCAE version 4.0. Grade 1 (>450 milliseconds [msec]), Grade 2 (>480 msec), Grade 3 (>500 msec). An increase is defined as an increase in CTCAE grade relative to Baseline grade. Data for any grade increase at worst case on therapy is presented.
Time Frame: Up to 2 years
Population: All Treated Population. Only those participants with data available at the indicated time points were analyzed. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Parts 1b and 1c as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 3 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants | 2 | 1 | 2 | 0 | 0 | 3 | 0 |  |  |  | 1 | 1 |  |  |

19. Primary Outcome: Part 2: Number of Participants With Any QTcF Interval Increases From Baseline According to Markedly Abnormal Criteria
Description: 12-lead ECG was planned to be performed to measure QTcF interval.
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Part 1: Objective Response Rate
Description: Objective response rate is defined as the percentage of participants achieving a confirmed best overall response of complete response (CR) or partial response (PR) evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1, where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeters (mm) in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Up to 47 months and 13 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Percentage of participants | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 |  |  |  | 0.0 | 33.3 |  |  |

21. Secondary Outcome: Part 2: Objective Response Rate
Description: Objective response rate is defined as the percentage of participants achieving a confirmed best overall response of CR or PR evaluated using RECIST v 1.1, where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Part 1: Disease Control Rate
Description: Disease control rate is defined as the percentage of participants with a confirmed best overall response of CR or PR or at least 12 weeks of stable disease per RECIST v 1.1.
Time Frame: Up to 47 months and 13 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Percentage of participants | 44.4 | 33.3 | 33.3 | 25.0 | 0.0 | 16.7 | 20.0 |  |  |  | 14.3 | 33.3 |  |  |

23. Secondary Outcome: Part 2: Disease Control Rate
Description: as for outcome 22
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Part 1: Time to Response
Description: Time to response is defined as the time from the date of first dose to the date of the first documented evidence of response (PR or CR).
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Parts 1b and 1c as no participants were enrolled. Values are presented based on the Kaplan-Meier analysis. Only participants with CR or PR are included in analysis. For arms with N=0, time to response could not be calculated as no participants had a confirmed CR or PR with in these arms.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Months | 5.6 [5.6 to 5.6] |  |  |  |  |  |  |  |  |  |  | 2.0 [1.6 to 2.4] |  |  |

25. Secondary Outcome: Part 2: Time to Response
Description: as for outcome 24
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Part 1: Duration of Response
Description: Duration of response is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause among participants who achieve an overall response (that is., a confirmed best overall response of CR or PR) by RECIST v 1.1.
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Parts 1b and 1c as no participants were enrolled. Values are presented based on the Kaplan-Meier analysis. Only participants with CR or PR are included in analysis. For arms with N=0, duration of response could not be calculated as no participants had a confirmed CR or PR with in these arms.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Months | 13.73 [13.73 to 13.73] |  |  |  |  |  |  |  |  |  |  | NA [16.82 to NA] — The final event experienced by participants within the treatment arm occurred in the first 50% of survival times. Hence, median and third-quartile could not be derived. |  |  |

27. Secondary Outcome: Part 2: Duration of Response
Description: as for outcome 26
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Part 1: Progression-free Survival
Description: Progression-free survival is defined as the interval of time (in months) between the date of first dose to the date of disease progression according to clinical or radiological assessment or death due to any causes, whichever occurs earliest. PFS was determined according to RECIST version 1.1. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Parts 1b and 1c as no participants were enrolled. Values are presented based on the Kaplan-Meier analysis. All participants (overall population) were included in analysis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Months | 2.79 [2.64 to 5.13] | 3.29 [2.46 to 3.61] | 2.60 [2.00 to 7.46] | 2.25 [1.45 to 3.96] | NA [NA to NA] — Progression-free Survival could not be calculated as no participants had an event in Part 1a: 250ng GSK1795091 + 24mg GSK3174998 arm. | 2.28 [1.91 to 2.79] | 1.41 [1.15 to 2.46] |  |  |  | 2.22 [1.91 to 2.43] | 2.37 [2.33 to 19.22] |  |  |

29. Secondary Outcome: Part 2: Progression-free Survival
Description: Progression-free survival is defined as the interval of time (in months) between the date of first dose to the date of disease progression according to clinical or radiological assessment or death due to any causes, whichever occurs earliest by RECIST v 1.1. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Part 1: Overall Survival
Description: Overall survival is defined as time from the date of first dose of study treatment (whichever investigational drug administered first) to the date of death due to any cause.
Time Frame: Up to 47 months and 13 days
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Months | 9.03 [6.29 to NA] — The final event experienced by participants within the treatment arm occurred in the first 75% of survival times. Hence, third-quartile could not be derived. | 7.75 [3.61 to 9.03] | 16.69 [8.03 to NA] — The final event experienced by participants within the treatment arm occurred in the first 75% of survival times. Hence, third-quartile could not be derived. | 6.72 [3.20 to 9.86] | 11.14 [11.14 to 11.14] | 4.48 [3.15 to 8.38] | 2.89 [2.37 to NA] — The final event experienced by participants within the treatment arm occurred in the first 75% of survival times. Hence, third-quartile could not be derived. |  |  |  | 3.91 [2.66 to NA] — The final event experienced by participants within the treatment arm occurred in the first 75% of survival times. Hence, third-quartile could not be derived. | NA [6.08 to NA] — The final event experienced by participants within the treatment arm occurred in the first 50% of survival times. Hence, median and third-quartile could not be derived. |  |  |

31. Secondary Outcome: Part 2: Overall Survival
Description: as for outcome 30
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

32. Secondary Outcome: Part 1a: Plasma Concentration of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of plasma concentration of GSK1795091. Pharmacokinetic (PK) Population consisted of all participants from the All Treated population for whom a PK sample was obtained, analyzed, measurable, and valid.
Time Frame: Day 1: Pre-dose, 10 minutes, 2, 4, 6, 24 hours; Day 8: Pre-dose, 10 minutes, 4 hours; Days 15 and 57: Pre-dose, 10 minutes, 4, 24 hours; Day 22: Pre-dose; Day 64: Pre-dose, 10 minutes; Days 78, 162, 246, 414 and 498: 10 minutes post-dose
Population: PK Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998
Number analyzed (Participants) | 9 | 5 | 9 | 4 | 2
Picogram per milliliter
  Day 1: Pre-dose, n=9,5,9,4,2 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  Day 1: 10 minutes, n=7,5,9,4,2: number analyzed (Participants) | 7 | 5 | 9 | 4 | 2
  Day 1: 10 minutes, n=7,5,9,4,2 | 3.960 [0.00 to 5.80] | 4.920 [4.00 to 11.90] | 28.800 [5.59 to 53.40] | 56.330 [43.60 to 68.05] | 82.175 [64.97 to 99.38]
  Day 1: 2 hours, n=8,5,9,4,2: number analyzed (Participants) | 8 | 5 | 9 | 4 | 2
  Day 1: 2 hours, n=8,5,9,4,2 | 1.580 [0.00 to 4.02] | 4.090 [2.49 to 5.92] | 29.200 [2.87 to 48.80] | 57.195 [35.97 to 63.79] | 62.285 [57.57 to 67.00]
  Day 1: 4 hours, n=8,5,9,4,2: number analyzed (Participants) | 8 | 5 | 9 | 4 | 2
  Day 1: 4 hours, n=8,5,9,4,2 | 3.680 [0.00 to 4.41] | 3.680 [2.29 to 5.67] | 27.300 [2.11 to 46.90] | 47.315 [33.66 to 61.52] | 60.945 [56.43 to 65.46]
  Day 1: 6 hours, n=8,3,9,4,1: number analyzed (Participants) | 8 | 3 | 9 | 4 | 1
  Day 1: 6 hours, n=8,3,9,4,1 | 0.000 [0.00 to 2.82] | 3.470 [2.50 to 4.66] | 25.700 [0.00 to 40.20] | 46.040 [32.61 to 64.30] | 57.180 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant.
  Day 1: 24 hours, n=8,5,9,4,2: number analyzed (Participants) | 8 | 5 | 9 | 4 | 2
  Day 1: 24 hours, n=8,5,9,4,2 | 0.000 [0.00 to 2.68] | 2.190 [0.00 to 3.70] | 15.800 [0.00 to 29.30] | 35.265 [27.09 to 44.10] | 39.120 [32.73 to 45.51]
  Day 8: Pre-dose, n=8,5,8,3,1: number analyzed (Participants) | 8 | 5 | 8 | 3 | 1
  Day 8: Pre-dose, n=8,5,8,3,1 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 5.25] | 4.590 [3.52 to 10.05] | 4.160 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant.
  Day 8: 10 minutes, n=9,5,8,3,1: number analyzed (Participants) | 9 | 5 | 8 | 3 | 1
  Day 8: 10 minutes, n=9,5,8,3,1 | 4.300 [0.00 to 10.20] | 6.160 [5.01 to 8.89] | 30.850 [2.28 to 60.54] | 71.910 [55.71 to 74.13] | 89.510 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant.
  Day 8: 4 hours, n=8,5,7,2,1: number analyzed (Participants) | 8 | 5 | 7 | 2 | 1
  Day 8: 4 hours, n=8,5,7,2,1 | 3.190 [0.00 to 6.80] | 3.790 [0.00 to 5.03] | 16.000 [0.00 to 37.40] | 61.830 [54.29 to 69.37] | 65.030 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant.
  Day 15: Pre-dose, n=9,3,9,2,0: number analyzed (Participants) | 9 | 3 | 9 | 2 | 0
  Day 15: Pre-dose, n=9,3,9,2,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 5.99] | 4.975 [4.73 to 5.22] |
  Day 15: 10 minutes, n=8,4,8,3,0: number analyzed (Participants) | 8 | 4 | 8 | 3 | 0
  Day 15: 10 minutes, n=8,4,8,3,0 | 5.255 [3.40 to 14.50] | 5.120 [4.35 to 8.96] | 35.625 [7.96 to 53.40] | 57.570 [46.52 to 76.81] |
  Day 15: 4 hours, n=9,3,6,3,0: number analyzed (Participants) | 9 | 3 | 6 | 3 | 0
  Day 15: 4 hours, n=9,3,6,3,0 | 2.830 [0.00 to 7.24] | 4.210 [2.75 to 5.02] | 25.675 [3.15 to 51.30] | 50.950 [43.71 to 62.64] |
  Day 15: 24 hours, n=9,3,8,3,0: number analyzed (Participants) | 9 | 3 | 8 | 3 | 0
  Day 15: 24 hours, n=9,3,8,3,0 | 0.000 [0.00 to 3.43] | 3.050 [2.36 to 3.43] | 18.970 [0.00 to 34.10] | 41.770 [36.87 to 50.89] |
  Day 22: Pre-dose, n=9,3,7,3,0: number analyzed (Participants) | 9 | 3 | 7 | 3 | 0
  Day 22: Pre-dose, n=9,3,7,3,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 5.60] | 4.450 [4.21 to 11.90] |
  Day 57: Pre-dose, n=6,3,6,0,0: number analyzed (Participants) | 6 | 3 | 6 | 0 | 0
  Day 57: Pre-dose, n=6,3,6,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 1.215 [0.00 to 24.77] |  |
  Day 57: 10 minutes, n=4,3,4,1,0: number analyzed (Participants) | 4 | 3 | 4 | 1 | 0
  Day 57: 10 minutes, n=4,3,4,1,0 | 6.400 [3.03 to 8.94] | 7.470 [6.08 to 18.20] | 32.600 [6.87 to 41.31] | 60.090 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |
  Day 57: 4 hours, n=4,3,6,1,0: number analyzed (Participants) | 4 | 3 | 6 | 1 | 0
  Day 57: 4 hours, n=4,3,6,1,0 | 3.855 [0.00 to 6.13] | 3.530 [3.36 to 16.30] | 13.735 [2.45 to 34.34] | 55.980 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |
  Day 57: 24 hours, n=6,4,6,2,0: number analyzed (Participants) | 6 | 4 | 6 | 2 | 0
  Day 57: 24 hours, n=6,4,6,2,0 | 0.000 [0.00 to 5.55] | 2.665 [2.41 to 11.60] | 16.595 [0.00 to 26.60] | 51.390 [45.48 to 57.30] |
  Day 64: Pre-dose, n=4,4,4,1,0: number analyzed (Participants) | 4 | 4 | 4 | 1 | 0
  Day 64: Pre-dose, n=4,4,4,1,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 3.040 [0.00 to 46.20] | 15.300 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |
  Day 64: 10 minutes, n=5,4,3,2,0: number analyzed (Participants) | 5 | 4 | 3 | 2 | 0
  Day 64: 10 minutes, n=5,4,3,2,0 | 3.340 [0.00 to 4.18] | 7.055 [4.95 to 20.60] | 26.700 [12.00 to 42.10] | 75.045 [74.38 to 75.71] |
  Day 78: 10 minutes, n=5,3,4,2,0: number analyzed (Participants) | 5 | 3 | 4 | 2 | 0
  Day 78: 10 minutes, n=5,3,4,2,0 | 3.980 [2.10 to 10.50] | 10.100 [6.80 to 24.80] | 22.700 [5.48 to 45.20] | 72.215 [67.82 to 76.61] |
  Day 162: 10 minutes, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 162: 10 minutes, n=1,0,0,0,0 | 3.450 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |  |
  Day 246: 10 minutes, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 246: 10 minutes, n=1,0,0,0,0 | 37.200 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |  |
  Day 414: 10 minutes, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 414: 10 minutes, n=1,0,0,0,0 | 18.600 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |  |
  Day 498: 10 minutes, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 498: 10 minutes, n=1,0,0,0,0 | 0.000 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |  |

33. Secondary Outcome: Part 1b: Plasma Concentration of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of plasma concentration of GSK1795091.
Time Frame: Day 1: Pre-dose, 10 minutes, 2, 4, 6, 24 hours; Day 8: Pre-dose, 10 minutes, 4 hours; Days 15 and 57: Pre-dose, 10 minutes, 4, 24 hours; Day 22: Pre-dose; Day 64: Pre-dose, 10 minutes; Day 78: 10 minutes post-dose
Population: PK Population. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Part 1b as no participants were enrolled. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609
Number analyzed (Participants) | 6 | 5 | 0 | 0 | 0
Picogram per milliliter
  Day 1: Pre-dose, n=6,5,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] |  |  |
  Day 1: 10 minutes, n=6,5,0,0,0 | 12.870 [0.00 to 15.80] | 32.300 [27.10 to 40.10] |  |  |
  Day 1: 2 hours, n=6,5,0,0,0 | 14.100 [0.00 to 28.80] | 29.770 [25.60 to 37.10] |  |  |
  Day 1: 4 hours, n=6,5,0,0,0 | 13.000 [0.00 to 14.40] | 25.330 [23.30 to 32.40] |  |  |
  Day 1: 6 hours, n=6,4,0,0,0: number analyzed (Participants) | 6 | 4 | 0 | 0 | 0
  Day 1: 6 hours, n=6,4,0,0,0 | 12.065 [0.00 to 13.40] | 23.690 [21.10 to 30.28] |  |  |
  Day 1: 24 hours, n=6,4,0,0,0: number analyzed (Participants) | 6 | 4 | 0 | 0 | 0
  Day 1: 24 hours, n=6,4,0,0,0 | 7.680 [0.00 to 9.17] | 19.650 [17.88 to 22.30] |  |  |
  Day 8: Pre-dose, n=5,4,0,0,0: number analyzed (Participants) | 5 | 4 | 0 | 0 | 0
  Day 8: Pre-dose, n=5,4,0,0,0 | 0.000 [0.00 to 0.00] | 2.215 [0.00 to 2.74] |  |  |
  Day 8: 10 minutes, n=5,4,0,0,0: number analyzed (Participants) | 5 | 4 | 0 | 0 | 0
  Day 8: 10 minutes, n=5,4,0,0,0 | 15.280 [2.97 to 17.28] | 29.550 [29.30 to 35.64] |  |  |
  Day 8: 4 hours, n=5,4,0,0,0: number analyzed (Participants) | 5 | 4 | 0 | 0 | 0
  Day 8: 4 hours, n=5,4,0,0,0 | 11.460 [0.00 to 15.94] | 23.850 [18.97 to 30.49] |  |  |
  Day 15: Pre-dose, n=4,3,0,0,0: number analyzed (Participants) | 4 | 3 | 0 | 0 | 0
  Day 15: Pre-dose, n=4,3,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 4.44] |  |  |
  Day 15: 10 minutes, n=4,4,0,0,0: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0
  Day 15: 10 minutes, n=4,4,0,0,0 | 16.000 [3.62 to 19.05] | 27.645 [25.70 to 49.04] |  |  |
  Day 15: 4 hours, n=4,4,0,0,0: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0
  Day 15: 4 hours, n=4,4,0,0,0 | 10.145 [2.70 to 15.20] | 24.100 [17.82 to 34.97] |  |  |
  Day 15: 24 hours, n=5,2,0,0,0: number analyzed (Participants) | 5 | 2 | 0 | 0 | 0
  Day 15: 24 hours, n=5,2,0,0,0 | 6.890 [0.00 to 12.48] | 14.735 [10.87 to 18.60] |  |  |
  Day 22: Pre-dose, n=5,2,0,0,0: number analyzed (Participants) | 5 | 2 | 0 | 0 | 0
  Day 22: Pre-dose, n=5,2,0,0,0 | 0.000 [0.00 to 2.45] | 1.015 [0.00 to 2.03] |  |  |
  Day 57: Pre-dose, n=3,1,0,0,0: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Day 57: Pre-dose, n=3,1,0,0,0 | 0.000 [0.00 to 3.33] | 2.300 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |
  Day 57: 10 minutes, n=3,2,0,0,0: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Day 57: 10 minutes, n=3,2,0,0,0 | 14.620 [12.20 to 17.86] | 28.155 [25.98 to 30.33] |  |  |
  Day 57: 4 hours, n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Day 57: 4 hours, n=1,1,0,0,0 | 12.140 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. | 25.510 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |
  Day 57: 24 hours, n=3,2,0,0,0: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Day 57: 24 hours, n=3,2,0,0,0 | 8.250 [6.59 to 11.44] | 17.530 [16.44 to 18.62] |  |  |
  Day 64: Pre-dose, n=1,2,0,0,0: number analyzed (Participants) | 1 | 2 | 0 | 0 | 0
  Day 64: Pre-dose, n=1,2,0,0,0 | 0.000 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. | 1.875 [0.00 to 3.75] |  |  |
  Day 64: 10 minutes, n=2,2,0,0,0: number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  Day 64: 10 minutes, n=2,2,0,0,0 | 6.910 [0.00 to 13.82] | 34.345 [32.14 to 36.55] |  |  |
  Day 78: 10 minutes, n=2,2,0,0,0: number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  Day 78: 10 minutes, n=2,2,0,0,0 | 6.980 [2.48 to 11.48] | 34.875 [32.02 to 37.73] |  |  |

34. Secondary Outcome: Part 1c: Plasma Concentration of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of plasma concentration of GSK1795091.
Time Frame: as for outcome 33
Population: PK Population. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Part 1c as no participants were enrolled. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 7 | 6 | 0 | 0 | 0
Picogram per milliliter
  Day 1: Pre-dose, n=7,6,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] |  |  |
  Day 1: 10 minutes, n=7,6,0,0,0 | 13.600 [0.00 to 14.00] | 27.965 [13.20 to 38.64] |  |  |
  Day 1: 2 hours, n=6,6,0,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0
  Day 1: 2 hours, n=6,6,0,0,0 | 11.475 [0.00 to 12.77] | 28.775 [10.50 to 56.63] |  |  |
  Day 1: 4 hours, n=7,6,0,0,0 | 9.890 [0.00 to 12.20] | 25.970 [10.10 to 32.63] |  |  |
  Day 1: 6 hours, n=7,6,0,0,0 | 9.460 [0.00 to 12.54] | 24.415 [8.83 to 33.69] |  |  |
  Day 1: 24 hours, n=7,6,0,0,0 | 8.370 [0.00 to 10.14] | 15.825 [6.31 to 24.03] |  |  |
  Day 8: Pre-dose, n=6,5,0,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0 | 0
  Day 8: Pre-dose, n=6,5,0,0,0 | 0.000 [0.00 to 0.00] | 2.060 [0.00 to 2.51] |  |  |
  Day 8: 10 minutes, n=7,5,0,0,0: number analyzed (Participants) | 7 | 5 | 0 | 0 | 0
  Day 8: 10 minutes, n=7,5,0,0,0 | 12.810 [0.00 to 16.00] | 24.260 [14.80 to 35.30] |  |  |
  Day 8: 4 hours, n=6,5,0,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0 | 0
  Day 8: 4 hours, n=6,5,0,0,0 | 9.420 [2.56 to 13.68] | 23.390 [12.30 to 27.70] |  |  |
  Day 15: Pre-dose, n=3,4,0,0,0: number analyzed (Participants) | 3 | 4 | 0 | 0 | 0
  Day 15: Pre-dose, n=3,4,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 3.26] |  |  |
  Day 15: 10 minutes, n=7,6,0,0,0 | 9.200 [0.00 to 14.70] | 28.015 [12.60 to 54.93] |  |  |
  Day 15: 4 hours, n=7,4,0,0,0: number analyzed (Participants) | 7 | 4 | 0 | 0 | 0
  Day 15: 4 hours, n=7,4,0,0,0 | 7.070 [0.00 to 11.60] | 17.825 [6.81 to 26.60] |  |  |
  Day 15: 24 hours, n=7,5,0,0,0: number analyzed (Participants) | 7 | 5 | 0 | 0 | 0
  Day 15: 24 hours, n=7,5,0,0,0 | 4.580 [0.00 to 8.42] | 11.230 [5.53 to 19.80] |  |  |
  Day 22: Pre-dose, n=4,3,0,0,0: number analyzed (Participants) | 4 | 3 | 0 | 0 | 0
  Day 22: Pre-dose, n=4,3,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 3.49] |  |  |
  Day 57: Pre-dose, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Day 57: Pre-dose, n=2,1,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |
  Day 57: 10 minutes, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Day 57: 10 minutes, n=2,1,0,0,0 | 14.665 [12.80 to 16.53] | 23.840 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |
  Day 57: 4 hours, n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Day 57: 4 hours, n=2,0,0,0,0 | 10.515 [10.13 to 10.90] |  |  |  |
  Day 57: 24 hours, n=2,2,0,0,0: number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  Day 57: 24 hours, n=2,2,0,0,0 | 7.460 [6.72 to 8.20] | 9.780 [4.87 to 14.69] |  |  |
  Day 64: Pre-dose, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Day 64: Pre-dose, n=2,1,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |
  Day 64: 10 minutes, n=3,1,0,0,0: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Day 64: 10 minutes, n=3,1,0,0,0 | 13.570 [11.50 to 14.00] | 31.680 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual plasma concentration for this single participant. |  |  |
  Day 78: 10 minutes, n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Day 78: 10 minutes, n=2,0,0,0,0 | 15.455 [14.71 to 16.20] |  |  |  |

35. Secondary Outcome: Part 1a: Maximum Plasma Concentration (Cmax) of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of Cmax of GSK1795091.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998
Number analyzed (Participants) | 9 | 5 | 9 | 4 | 2
Picogram per milliliter
  Day 1, n=7,5,9,4,2: number analyzed (Participants) | 7 | 5 | 9 | 4 | 2
  Day 1, n=7,5,9,4,2 | 4.180 [3.16 to 5.80] | 4.920 [4.00 to 11.9] | 29.20 [5.59 to 53.4] | 59.95 [43.6 to 68.1] | 82.18 [65.0 to 99.4]
  Day 8, n=8,5,8,3,1: number analyzed (Participants) | 8 | 5 | 8 | 3 | 1
  Day 8, n=8,5,8,3,1 | 4.720 [2.49 to 10.2] | 6.160 [5.01 to 8.89] | 30.85 [2.28 to 60.5] | 71.91 [55.7 to 74.1] | 89.51 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cmax for this single participant.
  Day 15, n=9,4,8,3,0: number analyzed (Participants) | 9 | 4 | 8 | 3 | 0
  Day 15, n=9,4,8,3,0 | 5.110 [2.47 to 14.5] | 5.120 [4.35 to 8.96] | 35.63 [7.96 to 53.4] | 57.57 [46.5 to 76.8] |
  Day 22, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 57, n=4,3,4,1,0: number analyzed (Participants) | 4 | 3 | 4 | 1 | 0
  Day 57, n=4,3,4,1,0 | 6.400 [3.03 to 8.94] | 7.470 [6.08 to 18.2] | 32.60 [6.87 to 41.3] | 60.09 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cmax for this single participant. |
  Day 64, n=5,4,3,2,0: number analyzed (Participants) | 5 | 4 | 3 | 2 | 0
  Day 64, n=5,4,3,2,0 | 3.340 [0.00 to 4.18] | 7.055 [4.95 to 20.6] | 26.70 [12.0 to 42.1] | 75.05 [74.4 to 75.7] |
  Day 78, n=5,3,4,2,0: number analyzed (Participants) | 5 | 3 | 4 | 2 | 0
  Day 78, n=5,3,4,2,0 | 3.980 [2.10 to 10.5] | 10.10 [6.80 to 24.8] | 22.70 [5.48 to 45.2] | 72.22 [67.8 to 76.6] |
  Day 162, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 162, n=1,0,0,0,0 | 3.450 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cmax for this single participant. |  |  |  |
  Day 246, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 246, n=1,0,0,0,0 | 37.20 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cmax for this single participant. |  |  |  |
  Day 414, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 414, n=1,0,0,0,0 | 18.60 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cmax for this single participant. |  |  |  |
  Day 498, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 498, n=1,0,0,0,0 | 0.000 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cmax for this single participant. |  |  |  |

36. Secondary Outcome: Part 1b: Cmax of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of Cmax of GSK1795091.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609
Number analyzed (Participants) | 6 | 5 | 0 | 0 | 0
Picogram per milliliter
  Day 1, n=6,5,0,0,0 | 14.95 [2.23 to 28.8] | 32.30 [27.1 to 40.1] |  |  |
  Day 8, n=5,4,0,0,0: number analyzed (Participants) | 5 | 4 | 0 | 0 | 0
  Day 8, n=5,4,0,0,0 | 15.28 [2.97 to 17.3] | 29.55 [29.3 to 35.6] |  |  |
  Day 15, n=4,4,0,0,0: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0
  Day 15, n=4,4,0,0,0 | 16.00 [3.62 to 19.1] | 27.80 [25.7 to 49.0] |  |  |
  Day 22, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 57, n=3,2,0,0,0: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Day 57, n=3,2,0,0,0 | 14.62 [13.2 to 17.9] | 28.16 [26.0 to 30.3] |  |  |
  Day 64, n=2,2,0,0,0: number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  Day 64, n=2,2,0,0,0 | 6.910 [0.00 to 13.8] | 34.35 [32.1 to 36.6] |  |  |
  Day 78, n=2,2,0,0,0: number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  Day 78, n=2,2,0,0,0 | 6.980 [2.48 to 11.5] | 34.88 [32.0 to 37.7] |  |  |

37. Secondary Outcome: Part 1c: Cmax of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of Cmax of GSK1795091.
Time Frame: as for outcome 33
Population: as for outcome 34
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0
Picogram per milliliter
  Day 1, n=6,6,0,0,0 | 13.75 [6.04 to 14.0] | 30.56 [13.2 to 56.6] |  |  |
  Day 8, n=6,5,0,0,0: number analyzed (Participants) | 6 | 5 | 0 | 0 | 0
  Day 8, n=6,5,0,0,0 | 13.53 [5.44 to 16.0] | 25.35 [14.8 to 35.3] |  |  |
  Day 15, n=6,6,0,0,0 | 10.19 [4.60 to 14.7] | 28.02 [12.6 to 54.9] |  |  |
  Day 22, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 57, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Day 57, n=2,1,0,0,0 | 14.67 [12.8 to 16.5] | 23.84 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cmax for this single participant. |  |  |
  Day 64, n=3,1,0,0,0: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Day 64, n=3,1,0,0,0 | 13.57 [11.5 to 14.0] | 31.68 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cmax for this single participant. |  |  |
  Day 78, n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Day 78, n=2,0,0,0,0 | 15.46 [14.7 to 16.2] |  |  |  |

38. Secondary Outcome: Part 1a: Area Under the Concentration-time Curve Over the Dosing Interval (AUC[0-tau]) GSK1795091
Description: Blood samples were collected at indicated time points for the determination of AUC(0-tau) of GSK1795091.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Full Range); unit: Hours*picogram per milliliter
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998
Number analyzed (Participants) | 5 | 5 | 8 | 3 | 1
Hours*picogram per milliliter
  Day 1, n=5,5,8,3,1 | 48.08 [35.0 to 276] | 227.6 [39.0 to 383] | 1804 [41.0 to 2540] | 3615 [2390 to 4300] | 4166 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual AUC(0-tau) for this single participant.
  Day 8, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 15, n=2,2,6,3,0: number analyzed (Participants) | 2 | 2 | 6 | 3 | 0
  Day 15, n=2,2,6,3,0 | 256.7 [191 to 322] | 318.3 [294 to 343] | 1907 [273 to 3000] | 3479 [3020 to 4900] |
  Day 22, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 57, n=0,3,2,1,0: number analyzed (Participants) | 0 | 3 | 2 | 1 | 0
  Day 57, n=0,3,2,1,0 |  | 267.9 [247 to 1140] | 2027 [1410 to 2640] | 3515 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual AUC(0-tau) for this single participant. |
  Day 64, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 78, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 162, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 246, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 414, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 498, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Part 1b: AUC(0-tau) GSK1795091
Description: Blood samples were collected at indicated time points for the determination of AUC(0-tau) of GSK1795091.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Median (Full Range); unit: Hours*picogram per milliliter
Arm/Group | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609
Number analyzed (Participants) | 4 | 4 | 0 | 0 | 0
Hours*picogram per milliliter
  Day 1, n=4,4,0,0,0 | 819.1 [721 to 899] | 1840 [1560 to 2120] |  |  |
  Day 8, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 15, n=3,2,0,0,0: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Day 15, n=3,2,0,0,0 | 661.9 [632 to 916] | 1453 [1100 to 1800] |  |  |
  Day 22, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 57, n=1,2,0,0,0: number analyzed (Participants) | 1 | 2 | 0 | 0 | 0
  Day 57, n=1,2,0,0,0 | 845.2 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual AUC(0-tau) for this single participant. | 1757 [1740 to 1780] |  |  |
  Day 64, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 78, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Part 1c: AUC(0-tau) GSK1795091
Description: Blood samples were collected at indicated time points for the determination of AUC(0-tau) of GSK1795091.
Time Frame: as for outcome 33
Population: as for outcome 34
Measure: Median (Full Range); unit: Hours*picogram per milliliter
Arm/Group | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 4 | 5 | 0 | 0 | 0
Hours*picogram per milliliter
  Day 1, n=4,5,0,0,0 | 851.7 [208 to 990] | 1611 [645 to 1710] |  |  |
  Day 8, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 15, n=3,2,0,0,0: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Day 15, n=3,2,0,0,0 | 566.9 [460 to 815] | 1189 [540 to 1840] |  |  |
  Day 22, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 57, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Day 57, n=2,1,0,0,0 | 778.0 [750 to 805] | 1640 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual AUC(0-tau) for this single participant. |  |  |
  Day 64, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 78, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Part 1a: Predose Concentration (Cpre) of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of Cpre of GSK1795091.
Time Frame: Days 1, 8, 15, 22, 57, 64, 78, 162, 246, 414 and 498: Pre-dose
Population: as for outcome 32
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998
Number analyzed (Participants) | 9 | 5 | 8 | 3 | 1
Picogram per milliliter
  Day 1, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 8, n=8,5,8,3,1: number analyzed (Participants) | 8 | 5 | 8 | 3 | 1
  Day 8, n=8,5,8,3,1 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 5.25] | 4.590 [3.52 to 10.1] | 4.160 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cpre for this single participant.
  Day 15, n=9,3,8,2,0: number analyzed (Participants) | 9 | 3 | 8 | 2 | 0
  Day 15, n=9,3,8,2,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 5.99] | 4.975 [4.73 to 5.22] |
  Day 22, n=9,3,7,3,0: number analyzed (Participants) | 9 | 3 | 7 | 3 | 0
  Day 22, n=9,3,7,3,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 5.60] | 4.450 [4.21 to 11.9] |
  Day 57, n=4,3,4,0,0: number analyzed (Participants) | 4 | 3 | 4 | 0 | 0
  Day 57, n=4,3,4,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 1.215 [0.00 to 6.02] |  |
  Day 64, n=4,4,4,1,0: number analyzed (Participants) | 4 | 4 | 4 | 1 | 0
  Day 64, n=4,4,4,1,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 3.040 [0.00 to 46.2] | 15.30 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cpre for this single participant. |
  Day 78, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 162, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 246, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 414, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 498, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Part 1b: Cpre of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of Cpre of GSK1795091.
Time Frame: Days 1, 8, 15, 22, 57, 64 and 78: Pre-dose
Population: as for outcome 33
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609
Number analyzed (Participants) | 5 | 4 | 0 | 0 | 0
Picogram per milliliter
  Day 1, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 8, n=5,4,0,0,0 | 0.000 [0.00 to 0.00] | 2.215 [0.00 to 2.74] |  |  |
  Day 15, n=4,3,0,0,0: number analyzed (Participants) | 4 | 3 | 0 | 0 | 0
  Day 15, n=4,3,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 4.44] |  |  |
  Day 22, n=5,2,0,0,0: number analyzed (Participants) | 5 | 2 | 0 | 0 | 0
  Day 22, n=5,2,0,0,0 | 0.000 [0.00 to 2.45] | 1.015 [0.00 to 2.03] |  |  |
  Day 57, n=3,1,0,0,0: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Day 57, n=3,1,0,0,0 | 0.000 [0.00 to 3.33] | 2.300 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cpre for this single participant. |  |  |
  Day 64, n=1,2,0,0,0: number analyzed (Participants) | 1 | 2 | 0 | 0 | 0
  Day 64, n=1,2,0,0,0 | 0.000 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cpre for this single participant. | 1.875 [0.00 to 3.75] |  |  |
  Day 78, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Part 1c: Cpre of GSK1795091
Description: Blood samples were collected at indicated time points for the determination of Cpre of GSK1795091.
Time Frame: Days 1, 8, 15, 22, 57, 64 and 78: Pre-dose
Population: as for outcome 34
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 5 | 5 | 0 | 0 | 0
Picogram per milliliter
  Day 1, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 8, n=5,5,0,0,0 | 0.000 [0.00 to 0.00] | 2.060 [0.00 to 2.51] |  |  |
  Day 15, n=3,4,0,0,0: number analyzed (Participants) | 3 | 4 | 0 | 0 | 0
  Day 15, n=3,4,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 3.26] |  |  |
  Day 22, n=3,3,0,0,0: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0
  Day 22, n=3,3,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 3.49] |  |  |
  Day 57, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Day 57, n=2,1,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cpre for this single participant. |  |  |
  Day 64, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Day 64, n=2,1,0,0,0 | 0.000 [0.00 to 0.00] | 0.000 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Cpre for this single participant. |  |  |
  Day 78, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Part 1a: Number of Participants With Present Antidrug Antibody (ADA) Against GSK3174998
Description: Serum samples were collected at indicated time points and tested for the presence of antibodies that bind to GSK3174998. The presence of anti-GSK3174998 antibodies were assessed using a titered approach using validated immunoassays (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 27 months
Population: All Treated Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998
Number analyzed (Participants) | 9 | 5 | 9 | 4 | 1
Participants | 5 | 0 | 2 | 1 | 0

45. Secondary Outcome: Part 1b: Number of Participants With the Present ADA Against GSK3359609
Description: Serum samples were collected at indicated time points and tested for the presence of antibodies that bind to GSK3359609. The presence of anti-GSK3359609 antibodies were assessed using a titered approach using validated immunoassays (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 27 months
Population: All Treated Population. Only those participants with data available at the indicated time points were analyzed. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Part 1b as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609
Number analyzed (Participants) | 4 | 3 | 0 | 0 | 0
Participants | 0 | 1 |  |  |

46. Secondary Outcome: Part 1c: Number of Participants With the Present ADA Against Pembrolizumab
Description: Serum samples were collected at indicated time points for the presence of antibodies that bind to pembrolizumab. The presence of anti-pembrolizumab antibodies were planned to be assessed using a titered approach using validated immunoassays (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 27 months
Population: All Treated Population. Data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Part 1c as no participants were enrolled. Samples were collected but will not be analyzed for the presence of anti-pembrolizumab antibodies as pembrolizumab immunogenicity has been previously characterized.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 7 | 6 | 0 | 0 | 0
Participants | NA — Samples were collected but will not be analyzed for the presence of anti-pembrolizumab antibodies as pembrolizumab immunogenicity has been previously characterized. | NA — Samples were collected but will not be analyzed for the presence of anti-pembrolizumab antibodies as pembrolizumab immunogenicity has been previously characterized. |  |  |

47. Secondary Outcome: Part 2a: Number of Participants With the Present ADA Against GSK3174998
Description: Serum samples were planned to be collected at indicated time points and tested for the presence of antibodies that bind to GSK3174998. The presence of anti-GSK3174998 antibodies were were planeed to be assessed using a titered approach using validated immunoassays (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998
Number analyzed (Participants) | 0

48. Secondary Outcome: Part 2b: Number of Participants With the Present ADA Against GSK3359609
Description: Serum samples were planned to be collected at indicated time points and tested for the presence of antibodies that bind to GSK3359609. The presence of anti-GSK3359609 antibodies were were planeed to be assessed using a titered approach using validated immunoassays (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2b: GSK1795091 + 80 mg GSK3359609
Number analyzed (Participants) | 0

49. Secondary Outcome: Part 2c: Number of Participants With the Present ADA Against Pembrolizumab
Description: Serum samples were planned to be collected at indicated time points and tested for the presence of antibodies that bind to pembrolizumab. The presence of anti-pembrolizumab antibodies were were planeed to be assessed using a titered approach using validated immunoassays (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0

50. Other Pre Specified Outcome: Part 1: Number of Participants With TEAEs and STEAEs Until End of the Study
Description: as for outcome 2
Time Frame: Up to 47 months and 13 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  TEAEs | 9 | 6 | 9 | 4 | 1 | 6 | 5 |  |  |  | 5 | 6 |  |  |
  STEAEs | 1 | 2 | 5 | 1 | 0 | 2 | 2 |  |  |  | 3 | 2 |  |  |

51. Other Pre Specified Outcome: Part 2: Number of Participants With TEAEs and STEAEs Until End of the Study
Description: as for outcome 2
Time Frame: Up to 47 months and 13 days
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

52. Other Pre Specified Outcome: Part 1: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: neutrophils (Neutro), lymphocytes (lympho) (Low), hemoglobin (Hb) (Low) and platelet count (PC). The laboratory parameters were graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Data for any worst-case on therapy any grade increase has been presented.
Time Frame: Up to 2 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  Neutro: n=8,6,9,4,2,6,4,0,0,0,6,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 4 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0
  Neutro: n=8,6,9,4,2,6,4,0,0,0,6,6,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 2 |  |  |
  Lympho (Low): n=8,6,9,4,2,6,4,0,0,0,6,6,0,0,0: number analyzed (Participants) | 8 | 6 | 9 | 4 | 2 | 6 | 4 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0
  Lympho (Low): n=8,6,9,4,2,6,4,0,0,0,6,6,0,0,0 | 7 | 3 | 4 | 0 | 0 | 5 | 0 |  |  |  | 2 | 3 |  |  |
  Hb (Low): n=9,6,9,4,2,6,4,0,0,0,7,6,0,0,0: number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 4 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Hb (Low): n=9,6,9,4,2,6,4,0,0,0,7,6,0,0,0 | 6 | 4 | 3 | 2 | 0 | 2 | 3 |  |  |  | 2 | 3 |  |  |
  PC: n=9,6,9,4,2,6,4,0,0,0,7,6,0,0,0: number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 4 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  PC: n=9,6,9,4,2,6,4,0,0,0,7,6,0,0,0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0 | 1 |  |  |

53. Other Pre Specified Outcome: Part 2: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: Blood samples were planned to be collected for the analysis of following hematology parameters: neutrophils (Neutro), lymphocytes (lympho), hemoglobin (Hb) and platelet count (PC).
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

54. Other Pre Specified Outcome: Part 1: Number of Participants With Worst-case Grade Change From Baseline in Chemistry Parameters
Description: Blood samples were collected for the analysis of following chemistry parameters: albumin (Hypo), ALP, ALT, AST, bilirubin, calcium (Hyper and Hypo), creatinine, glucose (Hyper and Hypo), potassium (Hyper and Hypo) and sodium (Hyper and Hypo). The laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Data for any worst-case on therapy any grade increase has been presented.
Time Frame: Up to 2 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1b: 150ng GSK1795091 + 80mg GSK3359609 | Part 1b: 200ng GSK1795091 + 80mg GSK3359609 | Part 1b: 250ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 150ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 200ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 250ng GSK1795091 + 200mg Pembrolizumab
Number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 6 | 5 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
Participants
  Albumin (Hypo): n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 4 | 2 | 2 | 2 | 0 | 2 | 2 |  |  |  | 1 | 3 |  |  |
  ALP: n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 5 | 1 | 4 | 1 | 0 | 3 | 2 |  |  |  | 2 | 1 |  |  |
  ALT: n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 2 | 4 | 2 | 0 | 3 | 2 |  |  |  | 1 | 2 |  |  |
  AST: n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 2 | 4 | 2 | 0 | 3 | 2 |  |  |  | 2 | 2 |  |  |
  Bilirubin: n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 0 | 2 | 0 | 0 | 1 | 1 |  |  |  | 2 | 1 |  |  |
  Calcium (Hyper): n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 |  |  |  | 1 | 2 |  |  |
  Calcium (Hypo): n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 |  |  |  | 2 | 0 |  |  |
  Creatinine: n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 4 | 3 | 1 | 2 | 0 | 2 | 1 |  |  |  | 0 | 1 |  |  |
  Glucose (Hyper): n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 7 | 0 | 4 | 2 | 2 | 3 | 1 |  |  |  | 1 | 3 |  |  |
  Glucose (Hypo): n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 |  |  |  | 0 | 1 |  |  |
  Potassium (Hyper): n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 1 | 0 | 3 | 0 | 0 | 3 | 0 |  |  |  | 0 | 2 |  |  |
  Potassium (Hypo): n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 4 | 0 | 0 | 0 | 1 | 1 | 0 |  |  |  | 2 | 2 |  |  |
  Sodium (Hyper): n=9,6,9,4,2,0,0,0,0,0,7,6,0,0,0: number analyzed (Participants) | 9 | 6 | 9 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 7 | 6 | 0 | 0 | 0
  Sodium (Hyper): n=9,6,9,4,2,0,0,0,0,0,7,6,0,0,0 | 0 | 0 | 1 | 0 | 0 |  |  |  |  |  | 0 | 1 |  |  |
  Sodium (Hypo): n=9,6,9,4,2,6,5,0,0,0,7,6,0,0,0 | 3 | 3 | 3 | 1 | 1 | 4 | 1 |  |  |  | 4 | 3 |  |  |

55. Other Pre Specified Outcome: Part 2: Number of Participants With Worst-case Grade Change From Baseline in Chemistry Parameters
Description: Blood samples were planned to be collected for the analysis of following chemistry parameters: albumin, ALP, ALT, AST, bilirubin, calcium, creatinine, glucose, potassium and sodium.
Time Frame: Up to 2 years
Population: All Treated Population. Data was not collected as no participants were enrolled in Part 2.
Arm/Group | Part 2a: GSK1795091 + 24 mg GSK3174998 | Part 2b: GSK1795091 + 80 mg GSK3359609 | Part 2c: GSK1795091 + 200 mg Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious TEAEs and STEAEs were collected up to 47 months and 13 days in Part 1
Description: All Treated Population. Data is presented for Part 1a of all arms, Part 1b and Part 1c (GSK1795091 50ng and 100mg arms only) as data was not collected for GSK1795091 150 ng, 200 ng and 250 ng arms of Parts 1b and 1c were not initiated as GSK1795091 was no longer supplied due to a manufacturing issue.
Arm/Group | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/9 | 5/6 | 4/9 | 4/4 | 1/2 | 5/6 | 3/5 | 4/7 | 3/6
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/6 | 5/9 | 1/4 | 0/2 | 2/6 | 2/5 | 3/7 | 2/6
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6 | 9/9 | 4/4 | 1/2 | 6/6 | 5/5 | 5/7 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 (N=9) | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 (N=6) | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 (N=9) | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 (N=4) | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 (N=2) | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 (N=6) | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 (N=5) | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab (N=7) | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a: 50ng GSK1795091 + 24mg GSK3174998 (N=9) | Part 1a: 100ng GSK1795091 + 24mg GSK3174998 (N=6) | Part 1a: 150ng GSK1795091 + 24mg GSK3174998 (N=9) | Part 1a: 200ng GSK1795091 + 24mg GSK3174998 (N=4) | Part 1a: 250ng GSK1795091 + 24mg GSK3174998 (N=2) | Part 1b: 50ng GSK1795091 + 80mg GSK3359609 (N=6) | Part 1b: 100ng GSK1795091 + 80mg GSK3359609 (N=5) | Part 1c: 50ng GSK1795091 + 200mg Pembrolizumab (N=7) | Part 1c: 100ng GSK1795091 + 200mg Pembrolizumab (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (5) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (11) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (4) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (10) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 5 (10) | 6 (20) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 2 (5)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (6) | 1 (2) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular microlithiasis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal reflux (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT03447314/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT03447314/SAP_001.pdf